CLINICAL TRIAL: NCT04400279
Title: COvid-19 Pandemic and Exercise (COPE) Trial: A Randomized Study Examining Physical Activities and Wellbeing in Individuals Mandated to Stay at Home
Brief Title: The COVID-19 Pandemic and Exercise Study
Acronym: COPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Eli Puterman, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H20-01497
Record Dates: First submitted 2020-05-21; First posted 2020-05-22 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Depressive Symptomatology; Psychological Distress; Health Behavior
Keywords: exercise; intervention; resilience; depression; general affect; flourishing; psychological distress
MeSH Terms: conditions — Health Behavior; Motor Activity; Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: PI will be blind to the allocation to the groups. Person sending out emails to participants to complete surveys will be blind to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Yoga Exercise group (Experimental): Using the Down Dog app, this group will be given access to an at-home personalized yoga practice, unique every time the participants complete it. Asked to complete yoga practice 4 times per week for 6 weeks. Weekly surveys will be administered to monitor wellbeing and health throughout the intervention. The second 6 weeks of the study, participants will have continued access to the Down Dog app and a final wellbeing and health survey will be administered at the end of the second 6 weeks.
  Interventions: Behavioral: Yoga group
- High Intensity Interval Training group (Experimental): Using the Down Dog app, this group will be given access to at-home bodyweight high intensity interval training (HIIT) workouts. Asked to complete these HIIT workouts 4 times per week for 6 weeks. Weekly surveys will be administered to monitor wellbeing and health throughout the intervention. The second 6 weeks of the study, participants will have continued access to the Down Dog app and a final wellbeing and health survey will be administered at the end of the second 6 weeks.
  Interventions: Behavioral: High Intensity Interval Training group
- Combination Yoga & HIIT group (Experimental): Using the Down Dog app, this group will be given access to both the unique yoga practice and bodyweight HIIT workouts. Asked to complete 2 yoga and 2 HIIT workouts per week. Weekly surveys will be administered to monitor wellbeing and health throughout the intervention. The second 6 weeks of the study, participants will have continued access to the Down Dog app and a final wellbeing and health survey will be administered at the end of the second 6 weeks.
  Interventions: Behavioral: Combination
- Control group (No Intervention): This group will be maintaining their pre-study activity levels for the first 6 weeks of the study. Weekly surveys will be administered to monitor wellbeing and health throughout the intervention. Then the participants will be given access to all the Down Dog apps (both yoga and HIIT included) to use as the participants please for the following 6 weeks. A final wellbeing and health survey at the end of the second 6 weeks will be administered.

INTERVENTIONS:
Behavioral: Yoga group — At-home yoga exercise instruction provided by a mobile/tablet app or through a computer web browser
  Arms: Yoga Exercise group
Behavioral: High Intensity Interval Training group — At-home HIIT exercise instruction provided by a mobile/tablet app or through a computer web browser
  Arms: High Intensity Interval Training group
Behavioral: Combination — At-home yoga & HIIT exercise instruction provided by a mobile/tablet app or through a computer web browser
  Arms: Combination Yoga & HIIT group

SUMMARY:
The COPE Trial is a randomized controlled trial that will provide currently isolated yet generally physically healthy 18-64 year old adults who are pre-retirement with the opportunity to receive a free 3-month subscription to either a yoga or moderate-to-high intensity aerobic exercise app or be randomized to a waitlist control group. Study outcomes include measures of psychological wellbeing and physical health.

DETAILED DESCRIPTION:
Global stay-at-home mandates implemented in response to the COVID-19 pandemic are having substantial negative effects on mental health. Developing approaches to maintain the mental health of all individuals during this unprecedented time of physical distancing is of paramount importance. In the proposed low cost randomized controlled trial (RCT), the investigators seek to answer whether the use of a mobile app that provides a variety of physical activities appropriate for home workouts [i.e., high intensity interval training (HIIT), yoga] can improve wellbeing and health in adults mandated to stay at home. Should the results of this trial support the efficacy of the intervention (via app delivery), this has the potential to be implemented and delivered rapidly and at scale.

Engaging in regular physical activity confers reduced risk for mental disorders (e.g. depression, anxiety) in clinical and non-clinical populations. The investigators' recent evidence also suggests that becoming physically active reduces depressive symptoms, as well as negative affect and rumination on a daily basis, while improving daily positive affect and a sense of control in highly stressed adults. With fitness centres currently closed by mandate, becoming physically active during the COVID-19 pandemic could prove to be a challenge for individuals who are typically inactive, those mandated to stay-at-home, or those who do not have opportunities to access outdoor spaces that provide the recommended two meters of distance between people. Thus, the investigators seek to support those living under stay-at-home mandates with access to mobile apps that provide opportunities to be physically active in the home environment.

The study will focus on physical activities requiring little physical space or equipment that are easily completed at home. The study includes yoga, a movement-based activity that promotes relaxation and mindfulness and only requires space for the full length and width of one's body, and a mat as equipment. Yoga has been shown to be effective in improving physical function and quality of life in RCTs. The study also includes whole body weight (WBW)-based HIIT, which also only requires a mat, making it an excellent home-based form of aerobic exercise. HIIT is characterized as bouts of high-intensity exercise combined with periods of recovery or lower intensity activity. Its physical and psychological benefits compared to continuous moderate intensity training are often evidenced to be equal or significantly stronger.

Aims. The primary outcome will be a measure of depressive symptomology. It is hypothesized that those who actively use the yoga and/or WBW-HIIT mobile apps will improve in their depressive symptomatology compared to the waitlist control group over the course of the 6-week RCT. The study will also include measures of, as secondary outcomes, psychological distress, quality of life, and self-reported physical health, and expect decreases in distress and increases in the remaining outcomes. The researchers will also investigate whether effects are stronger in those (a) who currently live alone vs. live with others, or (b) with poorer levels of psychological health pre-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-64
* Still working or pre-retirement
* Currently completing less than 150 minutes of moderate activity per week, and/or 75 minutes if vigorous activity per week
* has at-home internet/computer access
* English speaking

Exclusion Criteria:

* Retired
* Meeting activity guidelines (i.e. at least 150 min of moderate or 75 min of vigorous intensity exercise per week
* Major health conditions that limit ability to exercise
* Hospitalization in the last 3 months

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 334 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-11-28 (Actual); Study Completion 2020-11-28 (Actual)

PRIMARY OUTCOMES:
Changes in depressive symptomology over the course of the exercise intervention | Tracked weekly for 7 weeks (baseline, followed by 6 weeks of exercise intervention) and then a final CES-D survey at week 12
  The 10 Item Center for Epidemiologic Studies Depression Scale (CES-D) will be used in the baseline survey, and will be in each weekly survey to track changes in the CES-D over the study period. The possible range in scores is 0 to 30 depending on number of symptoms, with those symptoms weighted by frequency experienced in a week. Higher scores indicating more or more frequent symptoms.

SECONDARY OUTCOMES:
Changes in psychological stress as measured by the SCSQ over the course of the exercise intervention. | Tracked weekly for 7 weeks (baseline, followed by 6 weeks of exercise intervention) and then a final survey at week 12
  The 1 Item Statistics Canada Stress Question (SCSQ) will be used in the baseline survey and in each weekly survey to track changes in psychological stress over the study period. The SCSQ is a 1-item question with a possible scoring of 0 to 10, with higher scores indicating more stress.
Changes in psychological distress as measured by the K10 over the course of the exercise intervention. | Tracked weekly for 7 weeks (baseline, followed by 6 weeks of exercise intervention) and then a final survey at week 12
  The 10 Item Kessler Psychological Distress Scale (K10) will be used in the baseline survey and in each weekly survey to track changes in psychological distress over the study period. The K10 measures general psychological distress, typically over the last 30 days, but the investigators will be using the survey on a weekly basis to track changes potentially related to the exercise intervention. Scores range from 10-50, with higher scores indicating more symptoms or more frequent experience of those symptoms. Scores are weighted by how often the symptoms are experienced in a period of time, which in this case is the previous 7 days.
Changes in flourishing over the course of the exercise intervention | Tracked weekly for 7 weeks (baseline, followed by 6 weeks of exercise intervention) and then a final flourishing survey at week 12
  Diener's Flourishing scale will be used in the baseline survey, and will be in each weekly survey to track changes in flourishing over the study period. There are 8 items, phrased in a positive direction. Scores can range from 8 (strong disagreement with all items) to 56 (strong agreement with all items), with higher scores indicating individuals who have a more positive view of themselves in important areas of functioning.
Changes in resilience over the course of the exercise intervention | Tracked weekly for 7 weeks (baseline, followed by 6 weeks of exercise intervention) and then a final survey at week 12
  The Brief Resilience Scale (BRS) will be used in the baseline survey, and will be in each weekly survey to track changes in resilience over the study period. The BRS uses a mean scoring system with a possible range in scores from 1-5, higher scores indicate the individual perceives they have a better ability to 'bounce back' and recover from stressful events and/or situations.
Changes in life satisfaction over the course of the exercise intervention | Tracked weekly for 7 weeks (baseline, followed by 6 weeks of exercise intervention) and then a final survey at week 12
  A Life Satisfaction item, consisting of three questions, will be used in the baseline and weekly surveys to track changes over the study period. The first item is scored 0-10, with 10 indicating "the best possible life overall". Two follow-up questions asking individuals to rate their physical and mental/emotional health on a five point scale from poor to excellent. Higher scores overall indicate more satisfaction with life.
Changes in weekly strain as a result of health problems, financial/work issues, and relationship trouble using the Chronic Burden Scale over the course of the exercise intervention. | Tracked weekly for 7 weeks (baseline, followed by 6 weeks of exercise intervention) and then a final survey at week 12
  The Chronic Burden Scale (CBS) is an eight-item question asking about how much perceived strain individuals have experienced over the last week. This includes health problems with themselves, family members, and/or others close to them; problems with their job or ability to work; financial strain; and problems with relationships. There is a possible score of 8-32, with lower scores indicating less perceived strain.
Changes in general affect over the course of the exercise intervention | Tracked weekly for 7 weeks (baseline, followed by 6 weeks of exercise intervention) and then a final survey at week 12
  Using the positive and negative affect scale and a scale developed by Mroczek and Kolarz (1998) the investigators will be tracking participants affect. There are 25 items, scored 1 (felt all the time) to 5 (felt none of the time), with 13 negative affect and 18 positive affect items. PANAS Positive and negative affect will be considered separately, as will the positive items from Mroczek and Kolarz's measure, such that in each case higher scores will indicate higher amounts of positive or negative affect, respectively.
Changes in leisure time physical activity over the course of the exercise intervention | Tracked weekly for 7 weeks (baseline, followed by 6 weeks of exercise intervention) and then a final survey at week 12
  The investigators are tracking leisure time physical activity at baseline, and weekly (outside of the exercise intervention) using a version of the leisure score index (LSI) that was modified from the original LSI that was part of Godin's Leisure Time Exercise Questionnaire (GLTEQ). This question is open-ended and allows participants to tell us the frequency per week and time per exercise session of any mild, moderate, or strenuous exercise the participants have completed.
Changes in physical health symptomology over the course of the exercise intervention | Tracked weekly for 7 weeks (baseline, followed by 6 weeks of exercise intervention) and then a final survey at week 12
  A Physical Health item will be used in the baseline and weekly surveys to track changes in physical health (e.g. headache, backache, fever, sore throat, fatigue etc.) over the course of the study period. There are 13 physical symptoms, with the scoring based on how many symptoms were experienced in the past week. The scoring range is 0-13, with higher numbers indicating experiencing more negative physical health symptoms.
Changes in alcohol habits over the course of the exercise intervention | Tracked weekly for 7 weeks (baseline, followed by 6 weeks of exercise intervention) and then a final survey at week 12
  Using a 2-item alcohol habits question the investigators are tracking any changes in participants alcohol behaviours. Participants are asked if they drank at all in the last week, and if so, how many days per week they consumed alcohol. This is a modified version of the CDC's Behavioural Risk Factor Surveillance.
Tracking the amount of exercise variety participants feel they engage in | Tracked weekly for 7 weeks (baseline, followed by 6 weeks of exercise intervention) and then a final survey at week 12
  Using the Perceived Variety in Exercise (PVE) questionnaire, the investigators are tracking how varied participants feel their exercise activities are. There are 5 items asking about exercise variety, scored 1 (false) to 6 (true), with a possible score of 5-30; higher scores indicate greater perceived variety.

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification upon request and cleared for approval by principal investigator.
  All of the protocols, statistical analysis plan, informed consent form, analytic code.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 4 months following trial's end, materials will be made available. following publication, all data will be made available.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for the purpose for the purpose of meta-analyses and to achieve aims in the approved proposal. Investigators of the study need to approve the proposals. Proposals should be directed to eli.puterman@Ubc.ca
URL: https://osf.io/g9xqp

REFERENCES:
- [Background] Holmes EA, O'Connor RC, Perry VH, Tracey I, Wessely S, Arseneault L, Ballard C, Christensen H, Cohen Silver R, Everall I, Ford T, John A, Kabir T, King K, Madan I, Michie S, Przybylski AK, Shafran R, Sweeney A, Worthman CM, Yardley L, Cowan K, Cope C, Hotopf M, Bullmore E. Multidisciplinary research priorities for the COVID-19 pandemic: a call for action for mental health science. Lancet Psychiatry. 2020 Jun;7(6):547-560. doi: 10.1016/S2215-0366(20)30168-1. Epub 2020 Apr 15. PMID 32304649
- [Background] Pedersen BK, Saltin B. Exercise as medicine - evidence for prescribing exercise as therapy in 26 different chronic diseases. Scand J Med Sci Sports. 2015 Dec;25 Suppl 3:1-72. doi: 10.1111/sms.12581. PMID 26606383
- [Background] Stubbs B, Vancampfort D, Rosenbaum S, Firth J, Cosco T, Veronese N, Salum GA, Schuch FB. An examination of the anxiolytic effects of exercise for people with anxiety and stress-related disorders: A meta-analysis. Psychiatry Res. 2017 Mar;249:102-108. doi: 10.1016/j.psychres.2016.12.020. Epub 2017 Jan 6. PMID 28088704
- [Background] Schuch FB, Vancampfort D, Richards J, Rosenbaum S, Ward PB, Stubbs B. Exercise as a treatment for depression: A meta-analysis adjusting for publication bias. J Psychiatr Res. 2016 Jun;77:42-51. doi: 10.1016/j.jpsychires.2016.02.023. Epub 2016 Mar 4. PMID 26978184
- [Background] Hives BA, Buckler EJ, Weiss J, Schilf S, Johansen KL, Epel ES, Puterman E. The Effects of Aerobic Exercise on Psychological Functioning in Family Caregivers: Secondary Analyses of a Randomized Controlled Trial. Ann Behav Med. 2021 Feb 12;55(1):65-76. doi: 10.1093/abm/kaaa031. PMID 32421163
- [Background] Caplin A, Beauchamp MR, Weiss J, Schilf S, Hives B, DeLongis A, Johansen KL, Epel ES, Puterman E. Effects of Aerobic Exercise Training on Daily Psychological Processes in Family Caregivers: Secondary Analyses of a Randomized Controlled Trial. Affect Sci. 2021 Jan 28;2(1):48-57. doi: 10.1007/s42761-020-00026-6. eCollection 2021 Mar. PMID 36042918
- [Background] Sivaramakrishnan D, Fitzsimons C, Kelly P, Ludwig K, Mutrie N, Saunders DH, Baker G. The effects of yoga compared to active and inactive controls on physical function and health related quality of life in older adults- systematic review and meta-analysis of randomised controlled trials. Int J Behav Nutr Phys Act. 2019 Apr 5;16(1):33. doi: 10.1186/s12966-019-0789-2. PMID 30953508
- [Background] Buchheit M, Laursen PB. High-intensity interval training, solutions to the programming puzzle: Part I: cardiopulmonary emphasis. Sports Med. 2013 May;43(5):313-38. doi: 10.1007/s40279-013-0029-x. PMID 23539308
- [Background] Ramos JS, Dalleck LC, Tjonna AE, Beetham KS, Coombes JS. The impact of high-intensity interval training versus moderate-intensity continuous training on vascular function: a systematic review and meta-analysis. Sports Med. 2015 May;45(5):679-92. doi: 10.1007/s40279-015-0321-z. PMID 25771785
- [Background] Shepherd SO, Wilson OJ, Taylor AS, Thogersen-Ntoumani C, Adlan AM, Wagenmakers AJ, Shaw CS. Low-Volume High-Intensity Interval Training in a Gym Setting Improves Cardio-Metabolic and Psychological Health. PLoS One. 2015 Sep 24;10(9):e0139056. doi: 10.1371/journal.pone.0139056. eCollection 2015. PMID 26402859
- [Background] Andresen EM, Malmgren JA, Carter WB, Patrick DL. Screening for depression in well older adults: evaluation of a short form of the CES-D (Center for Epidemiologic Studies Depression Scale). Am J Prev Med. 1994 Mar-Apr;10(2):77-84. PMID 8037935
- [Background] Statistics (2012), Canada Canadian Community Health Survey. Share File, Knowledge Management and Reporting Branch, Ontario MOHLTC
- [Background] Kessler RC, Andrews G, Colpe LJ, Hiripi E, Mroczek DK, Normand SL, Walters EE, Zaslavsky AM. Short screening scales to monitor population prevalences and trends in non-specific psychological distress. Psychol Med. 2002 Aug;32(6):959-76. doi: 10.1017/s0033291702006074. PMID 12214795
- [Background] Diener, E., Wirtz, D., Tov, W., Kim-Prieto, C., Choi, D. W., Oishi, S., & Biswas-Diener, R. (2010). New well-being measures: Short scales to assess flourishing and positive and negative feelings. Social indicators research, 97(2), 143-156.
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Fleeson, W. (2004). The quality of American life at the end of the century. How healthy are we, 252-272.
- [Background] Cohen S, Schwartz JE, Epel E, Kirschbaum C, Sidney S, Seeman T. Socioeconomic status, race, and diurnal cortisol decline in the Coronary Artery Risk Development in Young Adults (CARDIA) Study. Psychosom Med. 2006 Jan-Feb;68(1):41-50. doi: 10.1097/01.psy.0000195967.51768.ea. PMID 16449410
- [Background] Watson, D., & Clark, L. A. (1999). The PANAS-X: Manual for the positive and negative affect schedule-expanded form.
- [Background] Mroczek DK, Kolarz CM. The effect of age on positive and negative affect: a developmental perspective on happiness. J Pers Soc Psychol. 1998 Nov;75(5):1333-49. doi: 10.1037//0022-3514.75.5.1333. PMID 9866191
- [Background] Courneya KS, Jones LW, Rhodes RE, Blanchard CM. Effects of different combinations of intensity categories on self-reported exercise. Res Q Exerc Sport. 2004 Dec;75(4):429-33. doi: 10.1080/02701367.2004.10609176. No abstract available. PMID 15673042
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Charles, S. T., & Almeida, D. M. (2006). Daily reports of symptoms and negative affect: Not all symptoms are the same. Psychology and Health, 21(1), 1-17.
- [Background] Centers for Disease Control and Prevention (CDC). (1984 - 2019). Behavioral Risk Factor Surveillance System Survey Questionnaire. Atlanta, Georgia: U.S. Department of Health and Human Services, Centers for Disease Control and Prevention.
- [Background] Sylvester BD, Standage M, Dowd AJ, Martin LJ, Sweet SN, Beauchamp MR. Perceived variety, psychological needs satisfaction and exercise-related well-being. Psychol Health. 2014;29(9):1044-61. doi: 10.1080/08870446.2014.907900. Epub 2014 Apr 22. PMID 24669787
- [Derived] Puterman E, Hives B, Mazara N, Grishin N, Webster J, Hutton S, Koehle MS, Liu Y, Beauchamp MR. COVID-19 Pandemic and Exercise (COPE) trial: a multigroup pragmatic randomised controlled trial examining effects of app-based at-home exercise programs on depressive symptoms. Br J Sports Med. 2022 May;56(10):546-552. doi: 10.1136/bjsports-2021-104379. Epub 2021 Sep 27. PMID 34580067